CLINICAL TRIAL: NCT00499993
Title: Phase III, Multicentre, Open Clinical Study on the Efficacy and Tolerability of a New Slow-release Formulation of Lanreotide (Autogel 120 mg) in Patients With Active Acromegaly
Brief Title: Efficacy and Tolerability of Lanreotide (Autogel 120 mg) in Patients With Acromegaly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-93-52030-077
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — lanreotide; Duration of Therapy

INTERVENTIONS:
Drug: lanreotide (Autogel formulation), duration of treatment 46-48 weeks

SUMMARY:
The purpose of the protocol, is to evaluate if lanreotide Autogel 120 mg is effective in the control of Growth Hormone (GH) secretion in patients with active acromegaly.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of active acromegaly, defined by serum GH levels above 5 µg/L, absence of reduction of serum GH levels below 1µg/L after oral glucose tolerance test (OGTT) and abnormal IGF-1 values

Exclusion Criteria:

* Patients who have undergone pituitary surgery less than 3 months before selection
* Patients previously treated with radiotherapy
* Patients previously treated with somatostatin analogue except for a pre-surgical treatment not longer than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2001-01; Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Growth hormone assessment | At every visit

SECONDARY OUTCOMES:
Insulin-like Growth Factor 1 (IGF-1) and Acid-Labile Subunit (ALS) assessments | At every visit (with the exception of ALS at study inclusion)
Prolactin (PRL) assessment | At study inclusion, visit 1 and at the final visit of the study
Lanreotide assessment | At every visit
Clinical symptoms | At every visit
Quality of life | At visit 1 and at the final visit of the study
Tumour size | At inclusion and at the final visit of the study
Evaluation of carotid vessels (on an optional basis) | At inclusion and at the final visit of the study
Safety assessment evaluated by clinical data | At every visit
Safety assessment evaluated by laboratory data | At inclusion visit and at the final visit of the study

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (24):
- Italy (24):
  - Ospedali Riuniti di Bergamo, Bergamo
  - Ospedale Maggiore, Bologna
  - Clinica Medica - Sezione II Medicina Endocrinologia, Brescia
  - Università deglis Studi di Cagliari, Cagliari
  - Ospedale Garibaldi, Catania
  - Università degli Studi di Ferrara, Ferrara
  - Università degli Studi di Firenze, Florence
  - D.i.S.E.M. Dipartimento di Scienze Endocrinologiche e Metaboliche, Genova
  - Istituto Auxologico, Milan
  - Ospedale Maggiore IRCCS, Milan
  - Ospedale di Niguarda Cà Granda, Milan
  - Università "Federico II" di Napoli, Napoli
  - Ospedale "S. Luigi Gonzaga", Orbassano (TO)
  - Università degli Studi di Padova, Padua
  - Azienda Ospedaliera "V. Cervello", Palermo
  - Ospedale Cisanello, Pisa
  - Servizio di Endocrinologia, Reggio Emilia
  - Università "La Sapienza" di Roma, Roma
  - Policlinico Agostino Gemelli, Roma
  - Istituto di Patologia Speciale Medica e Metodologia Clinica, Sassari
  - Università degli Studi di Ancona, Ospedale Umberto I, Sede Di Torrette (AN) Ancona
  - Ospedale Molinette, Torino
  - Ospedale Cà Foncello, Treviso
  - Ospedale Santa Maria della Misericordia, Udine

REFERENCES:
- [Result] Lombardi G, Minuto F, Tamburrano G, Ambrosio MR, Arnaldi G, Arosio M, Chiarini V, Cozzi R, Grottoli S, Mantero F, Bogazzi F, Terzolo M, Tita P, Boscani PF, Colao A. Efficacy of the new long-acting formulation of lanreotide (lanreotide Autogel) in somatostatin analogue-naive patients with acromegaly. J Endocrinol Invest. 2009 Mar;32(3):202-9. doi: 10.1007/BF03346453. PMID 19542735